CLINICAL TRIAL: NCT02539862
Title: Pilot Study Evaluating the Efficacy of the Management of an Online Program of Cognitive Behavioral Therapy for Primary Insomnia
Brief Title: Evaluating the Efficacy of the Management of an Online Program of Cognitive Behavioral Therapy for Primary Insomnia
Acronym: NEXPERTSANTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9454
Record Dates: First submitted 2015-07-24; First posted 2015-09-03 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; behavioral and cognitive therapies
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive behavioral therapy online (Experimental): patients receive cognitive behavioral therapy via an online program
  Interventions: Other: cognitive behavioral therapy online
- no cognitive behavioral therapy online (Other): patients receive psychoeducation by a doctor
  Interventions: Other: psychoeducation

INTERVENTIONS:
Other: cognitive behavioral therapy online — The cognitive behavioral therapy online program is delivered through an accessible web application on a web browser with a personal password
  Arms: cognitive behavioral therapy online
Other: psychoeducation — the psychoeducation is delivered by a doctor
  Arms: no cognitive behavioral therapy online

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the management of chronic primary insomnia patients by a computer program guidance of behavioral and cognitive therapies for insomnia (BCT-I).

DETAILED DESCRIPTION:
Chronic insomnia is a common sleep disorder (prevalence = 10%) and a risk identified on the physical and mental health. Currently, the treatment involves the prescription of drug treatments by general practitioners, which may be unsuitable for the medium term. It is better to turn to Behavioral and Cognitive Therapies for Insomnia (BCT-I) in the case of primary chronic insomnia. The objective of this study is to evaluate the effectiveness of a computer program guidance BCT-I in patients with chronic primary insomnia. This biomedical research psychotherapeutic assessment will be randomized, controlled versus psychoeducation and conducted in 46 patients with chronic primary insomnia (defined according to Diagnostic and Statistical Manual-5) for which a supported by BCT-I is indicated.

The 46 patients will be randomized into two groups. The subjects in Group 1 will be supported by BCT-I online. And the subjects in group 2 will receive psychoeducation. All patients will be followed by the research team for three months, during which 3 visits (V0 = pre-selection; V1 = visit of randomization and start of the program; V2 = 3 months follow-up visit and end of the study) will be performed in the University Hospital Sleep Disorder Unit of Montpellier. Patients in Group 1 will conduct BCT-I online at home therapy. Patients in group 2 will receive a structured 45-minute session information insomnia (psychoeducation = work performed daily by clinicians in charge of insomnia problems) to the visit 1. All patients in the study will be equipped 2 sensors for the registration of sleep data.

The primary endpoint will be based on the severity of insomnia measured by the ISI after the last online psychotherapy session (3 months) between the 2 groups of patients (BCT-I online and without treatment - psychoeducation ). The analyse efficacity to be conducted by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 65
* disorder diagnosis of chronic insomnia (according to Diagnostic and Statistical Manual-5)
* sleep efficiency <80%
* Index severe insomnia: ISI> 14/28
* have a computer at home
* Practicing internet regularly in everyday life
* have a personal email address

Exclusion Criteria:

* Clinically suffer from insomnia comorbid linked to other sleep disorders
* Presenting an unbalanced psychiatric disorder
* Have Score Beck Depression Inventory (BDI-II) >29
* Have neurological disorders
* Have severe medical conditions that can affect the quality of sleep
* Have Hypnotic, Anxiolytic, antidepressants Treatment > 2
* Have antipsychotics, opioids, anticonvulsants, anti-parkinson treatment
* Having a disorder of substance use (alcohol, drugs) in the last 6 months
* Having undertaken a meridian trance journey (± 3H) in the preceding month or during the study period
* Already be treated with CBT-I

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
insomnia severity measured | 100 days
  The primary endpoint will focus on the severity of insomnia measured by the Index severe insomnia (ISI) at the end of the last session of CBT (3 months) between the 2 groups of patients (CBT-I online and psychoeducation).

SECONDARY OUTCOMES:
sleep efficiency | 100 days
  duration of of sleep time compared to the time window passed to bed
Sleep latency | 100 days
  collection of data with actiwatch2 sensor
duration of night wakings | 100 days
  collection of data with actiwatch2 sensor
total sleep time | 100 days
  The total sleep time measured by sleep diary and actometer (Actiwatch 2 Sleep).
Sleep quality | 100 days
  sleepiness score assessed by a specific questionnaire
quantity of hypnotic treatment | 100 days
  number of hypnotic which will be consume by patient
adherence to CBT-I program online | 100 days
  the number of steps performed in the program, and the weekly frequency of connection.

CONTACTS AND LOCATIONS:
Overall Officials: Dauvilliers Yves, Principal Investigator — Unit of sleep disorders

REFERENCES:
- [Background] Leger D, Levy E, Paillard M. The direct costs of insomnia in France. Sleep. 1999 May 1;22 Suppl 2:S394-401. PMID 10394613
- [Background] Leigh JP. Employee and job attributes as predictors of absenteeism in a national sample of workers: the importance of health and dangerous working conditions. Soc Sci Med. 1991;33(2):127-37. doi: 10.1016/0277-9536(91)90173-a. PMID 1887276
- [Background] Morin CM, Culbert JP, Schwartz SM. Nonpharmacological interventions for insomnia: a meta-analysis of treatment efficacy. Am J Psychiatry. 1994 Aug;151(8):1172-80. doi: 10.1176/ajp.151.8.1172. PMID 8037252
- [Background] Murtagh DR, Greenwood KM. Identifying effective psychological treatments for insomnia: a meta-analysis. J Consult Clin Psychol. 1995 Feb;63(1):79-89. doi: 10.1037//0022-006x.63.1.79. PMID 7896994
- [Background] Gagnon C, Belanger L, Ivers H, Morin CM. Validation of the Insomnia Severity Index in primary care. J Am Board Fam Med. 2013 Nov-Dec;26(6):701-10. doi: 10.3122/jabfm.2013.06.130064. PMID 24204066
- [Background] Smith MT, Perlis ML, Park A, Smith MS, Pennington J, Giles DE, Buysse DJ. Comparative meta-analysis of pharmacotherapy and behavior therapy for persistent insomnia. Am J Psychiatry. 2002 Jan;159(1):5-11. doi: 10.1176/appi.ajp.159.1.5. PMID 11772681
- [Background] Irwin MR, Cole JC, Nicassio PM. Comparative meta-analysis of behavioral interventions for insomnia and their efficacy in middle-aged adults and in older adults 55+ years of age. Health Psychol. 2006 Jan;25(1):3-14. doi: 10.1037/0278-6133.25.1.3. PMID 16448292
- [Background] I. Okajima, Y. Komada, and Y. Inoue, A meta-analysis on the treatment effectiveness of cognitive behavioral therapy for primary insomnia. Sleep and Biological Rhythms, 2011. 9(1): p. 24-34.
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Ritterband LM, Thorndike FP, Gonder-Frederick LA, Magee JC, Bailey ET, Saylor DK, Morin CM. Efficacy of an Internet-based behavioral intervention for adults with insomnia. Arch Gen Psychiatry. 2009 Jul;66(7):692-8. doi: 10.1001/archgenpsychiatry.2009.66. PMID 19581560
- [Background] Morin CM, Bootzin RR, Buysse DJ, Edinger JD, Espie CA, Lichstein KL. Psychological and behavioral treatment of insomnia:update of the recent evidence (1998-2004). Sleep. 2006 Nov;29(11):1398-414. doi: 10.1093/sleep/29.11.1398. PMID 17162986
- [Background] NIH State-of-the-Science Conference Statement on manifestations and management of chronic insomnia in adults. NIH Consens State Sci Statements. 2005 Jun 13-15;22(2):1-30. PMID 17308547
- [Background] Schutte-Rodin S, Broch L, Buysse D, Dorsey C, Sateia M. Clinical guideline for the evaluation and management of chronic insomnia in adults. J Clin Sleep Med. 2008 Oct 15;4(5):487-504. PMID 18853708
- [Background] Thorndike FP, Ritterband LM, Gonder-Frederick LA, Lord HR, Ingersoll KS, Morin CM. A randomized controlled trial of an internet intervention for adults with insomnia: effects on comorbid psychological and fatigue symptoms. J Clin Psychol. 2013 Oct;69(10):1078-93. doi: 10.1002/jclp.22032. Epub 2013 Aug 28. PMID 24014057
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Chevalier J, de Pouvourville G. Valuing EQ-5D using time trade-off in France. Eur J Health Econ. 2013 Feb;14(1):57-66. doi: 10.1007/s10198-011-0351-x. Epub 2011 Sep 21. PMID 21935715
- [Background] Leger D, Morin CM, Uchiyama M, Hakimi Z, Cure S, Walsh JK. Chronic insomnia, quality-of-life, and utility scores: comparison with good sleepers in a cross-sectional international survey. Sleep Med. 2012 Jan;13(1):43-51. doi: 10.1016/j.sleep.2011.03.020. Epub 2011 Nov 16. PMID 22093806
- [Background] Cartwright RD. Alcohol and NREM parasomnias: evidence versus opinions in the international classification of sleep disorders, 3rd edition. J Clin Sleep Med. 2014 Sep 15;10(9):1039-40. doi: 10.5664/jcsm.4050. No abstract available. PMID 25221449